CLINICAL TRIAL: NCT06928142
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Sibeprenlimab Administered Subcutaneously in Participants With Sjögren's
Brief Title: A Trial to Evaluate the Efficacy and Safety of Sibeprenlimab Administered Subcutaneously in Participants With Sjögren's
Acronym: EnVISage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 417-201-00042
Record Dates: First submitted 2025-03-25; First posted 2025-04-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sjogren Disease
Keywords: Sibeprenlimab; Autoimmune Diseases; Immune System Diseases; Dry Mouth; Dry Eyes; Salivary Gland Disorders; Lacrimal Gland Disorders; Immunoglobulin G; EnVISage
MeSH Terms: conditions — Autoimmune Diseases; Immune System Diseases; Xerostomia; Dry Eye Syndromes; Salivary Gland Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 400 mg Sibeprenlimab (Experimental)
  Interventions: Biological: Sibeprenlimab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sibeprenlimab — 400 mg administered SC Q4 weeks
  Arms: 400 mg Sibeprenlimab
Other: Placebo — Administered SC Q4 weeks
  Arms: Placebo

SUMMARY:
This is a phase 2 study to evaluate the effects of sibeprenlimab 400 mg administered subcutaneously (SC) every 4 (Q4) weeks as an add-on to background treatment in participants with Sjögren's disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, proof-of-concept study followed by an optional open-label extension to evaluate the efficacy and safety of sibeprenlimab 400 mg administered SC Q4 weeks as an add-on to background treatment in participants with Sjögren's disease.

The primary objective is to compare the effect of sibeprenlimab versus placebo added to background treatment on European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) scores at 28 weeks.

The key secondary objective is to compare the effect of sibeprenlimab versus placebo added to background treatment on European League Against Rheumatism Sjögren's Syndrome Patient-Reported Index (ESSPRI) at 28 weeks.

Approximately 80 participants who have a diagnosis of Sjögren's disease according to the 2016 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria will be randomized with approximately 40 participants in the sibeprenlimab group and 40 participants in the placebo group.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with Sjögren's disease.
* ESSDAI score (which measures disease activity) must be 5 or higher.
* Salivary flow rate must be at least 0.05 mL/min.
* Serum IgG level must be higher than 900 mg/dL.
* Must be able to communicate well with the investigator and agree to follow the trial requirements.
* Participants can continue certain medications (hydroxychloroquine, methotrexate, leflunomide, or azathioprine) if they have been on a stable dose for at least 30 days.
* Corticosteroid dose must be stable and no more than 10 mg/day for at least 30 days.
* Test positive for anti-Ro52 and/or anti-Ro60 antibodies.

Key Exclusion Criteria:

* Another active autoimmune rheumatic disease.
* Prior use of B-cell depleting therapy or prohibited immunosuppressants.
* Significant comorbidities including uncontrolled type 2 diabetes, malignancy, and chronic and/or acute infections.
* Suicidal ideation or behavior based on the Patient Health Questionnaire-9 (PHQ-9).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) score | 28 weeks
  Higher scores on the ESSDAI indicate a worse outcome, as they reflect higher disease activity. Minimum value is 0 and the maximum value is 123.

SECONDARY OUTCOMES:
Change from baseline in European League Against Rheumatism Sjögren's Syndrome Patient-Reported Index (ESSPRI) score | 28 weeks
  Higher scores on the ESSPRI indicate a worse outcome, as they reflect higher levels of patient-reported symptoms. Minimum value is 0, maximum value is 10.
Incidence of treatment-emergent adverse events (TEAEs) | 28 weeks
Incidence of treatment-emergent adverse events (TEAEs) by National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade | 28 weeks
Incidence of treatment-emergent adverse events (TEAEs) with an outcome of death | 28 weeks
Incidence of serious treatment-emergent adverse events (TEAEs) | 28 weeks
Incidence of treatment-emergent adverse events (TEAEs) leading to discontinuation of the investigational medicinal product (IMP) | 28 weeks
Proportion of participants with minimal clinical improvement defined as European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) reduction ≥ 3 points from baseline | At 28 weeks
  Higher scores on the ESSDAI indicate a worse outcome, as they reflect higher disease activity. Minimum value is 0 and the maximum value is 123.
Proportion of participants with minimal clinical improvement defined as European League Against Rheumatism Sjögren's Syndrome Patient-Reported Index (ESSPRI) reduction ≥ 1 point from baseline | At 28 weeks
  Higher scores on the ESSPRI indicate a worse outcome, as they reflect higher levels of patient-reported symptoms. Minimum value is 0, maximum value is 10.
Change from baseline in individual European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) domains | At 28 weeks
  Higher scores on the ESSDAI indicate a worse outcome, as they reflect higher disease activity. Minimum value is 0 and the maximum value is 123.
Change from baseline in salivary flow rate | At 28 weeks
Change from baseline in tear flow rate | At 28 weeks
Change from baseline in Clinical European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ClinESSDAI) score | At 28 weeks
  Higher scores on the ClinESSDAI indicate a worse outcome, as they reflect higher disease activity. Minimum value is 0 and the maximum value is 123.
Change from baseline in Physician Global Assessment (PhGA) score | At 28 weeks
  Higher scores on the PhGA indicate a worse outcome, as they reflect a higher assessment of disease activity or severity by the physician. Minimum value is 0 and the maximum value is 10.
Change from baseline in Patient Global Assessment (PaGA) score of participant outcomes | At 28 weeks
  Higher scores on the PaGA indicate a worse outcome, as they reflect a higher assessment of disease severity or impact by the patient. Minimum value is 0 and the maximum value is 10.
Change from baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) score | At 28 weeks
  Higher FACIT-Fatigue scores indicate a better outcome, as they reflect less fatigue. Minimum value is 0 and the maximum value is 52.
Change from baseline in 36 Item Short-Form Survey Version 2 (SF-36v2) Physical Component Summary Scale score and Mental Component Summary Scale score | At 28 weeks
  Higher scores on the SF-36v2 indicate a better outcome, as they reflect better health status and quality of life. Minimum value is 0 and the maximum value is 100.
Change from baseline in patient-reported Sjögren's disease diary score | At 28 weeks
  Higher diary score indicates more severe symptoms and greater impact on the patient's daily life. Minimum value is 0 and the maximum value is 10.
Proportion of participants with minimal clinical improvement, defined as Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) score increase of ≥ 4 from baseline | At 28 weeks
  Higher FACIT-Fatigue scores indicate a better outcome, as they reflect less fatigue. Minimum value is 0 and the maximum value is 52.
Time to the first occurrence of minimal clinical improvement in ESSDAI | Week 28
Time to the first occurrence of minimal clinical improvement in ESSPRI | Week 28
Percent change from baseline in total serum IgA | Week 28
Percent change from baseline in total serum IgG | Week 28
Percent change from baseline in total serum IgM | Week 28
Percent change from baseline in total serum free APRIL (a proliferation-inducing ligand) concentrations | Week 28
Cmax of sibeprenlimab | 28 weeks
Tmax of sibeprenlimab | 28 weeks
Area Under the Curve (AUC) of sibeprenlimab | 28 weeks
Serum concentration of sibeprenlimab | 28 weeks
Presence or absence of serum antidrug antibody (ADA) to sibeprenlimiab | 28 weeks

CONTACTS AND LOCATIONS:
Locations (73):
- United States (23):
  - Medvin Clinical Research - Riverside, Riverside, California
  - Medvin Clinical Research - Tujunga, Tujunga, California
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Clinical Research of West Florida Inc, Clearwater, Florida
  - GNP Research - Florida, Cooper City, Florida
  - Vantage Clinical Trials - Tampa - ClinEdge - PPDS, Tampa, Florida
  - OrthoIllinois, LTD, Rockford, Illinois
  - Arnold Arthritis and Rheumatology, Skokie, Illinois
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - Kirk Kerkorian School of Medicine UNLV, Las Vegas, Nevada
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Bradenton Research Center Inc, The Bronx, New York
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - Ruppert Health Center, Toledo, Ohio
  - STAT Research, Vandalia, Ohio
  - Toyos Clinic-Memphis, Nashville, Tennessee
  - Allen Arthritis, Allen, Texas
  - Tekton Research, LLC, Austin, Texas
  - Advanced Rheumatology of Houston, Houston, Texas
  - Accurate Clinical Research - Houston, Houston, Texas
  - Accurate Clinical Management, LLC, Katy, Texas
  - R & H Clinical Research, Katy, Texas
- Argentina (10):
  - Consultorios Médicos Dr. Doreski - Fundacion Respirar - PPDS, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto CER S.A., Quilmes, Buenos Aires
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario, Santa Fe Province
  - Clínica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán, Tucumán Province
  - DOM Centro de Reumatología, Buenos Aires
  - Expertia S.A- Mautalén Salud e Investigación, Buenos Aires
  - Maffei Centro Médico, Buenos Aires
  - Aprillus Asistencia e Investigacion de Arcis Salud SRL, Buenos Aires
  - Centro Polivalente de Asistencia e Investigación Clínica - CER San Juan, San Juan
- Bulgaria (5):
  - Medical Center Medconsult Pleven OOD, Pleven
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD-15 A Vassil Aprilov Boulevard, Plovdiv
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Diagnostic- Consultative Center Convex EOOD, Sofia
  - Medical Center- Nova Clinic, Varna
- Germany (4):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Mvz Rheumatologie Und Autoimmunmedizin Hamburg Gmbh, Hamburg
  - Medicover München Ost MVZ, München
- Greece (4):
  - Olympion General Clinic, Pátrai, Achaïa
  - Laiko General Hospital of Athens (Site 1), Athens, Attica
  - Laiko General Hospital of Athens (Site 2), Athens, Attica
  - General Hospital ''Asklepieio Voulas'', Voula, Attica
- Mexico (4):
  - Mediadvance Clinical S.A.P.I. de C.V, San Felipe, Chihuahua
  - Centro de Estudios de Investigacion Basica Y Clinica SC, Guadalajara, Jalisco
  - PanAmerican Clinical Research - Domingo Sarmiento 2784 - PPDS, Zapopan, Jalisco
  - Centro de Investigación y Tratamiento Reumatológico S.C, Mexico City, Mexico City
- Poland (14):
  - Twoja Przychodnia PCM, Poznan, Greater Poland Voivodeship
  - Med-Polonia Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Prywatna Praktyka Lekarska Pawel Hrycaj, Poznan, Greater Poland Voivodeship
  - Pracownia Badan Klinicznych Salus - ul. Ołtaszyńska 92c/3, Wroclaw, Lower Silesian Voivodeship
  - ETG Siedlce - PPDS, Siedlce, Masovian Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Dr hab. Med. Eleonory Reicher, Warsaw, Masovian Voivodeship
  - Klinika Reuma Park sp . zoo Sp.k., Warsaw, Masovian Voivodeship
  - Centrum Medyczne K2J2 - Wołomin, Wołomin, Masovian Voivodeship
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - NZOZ Holsamed - Oddzial Libero, Katowice
  - Zespol Poradni Specjalistycznych REUMED- Wallenroda 2F/4, Lublin
  - Pratia Poznan - PPDS, Poznan
  - ETG Warszawa - PPDS, Warsaw
- Romania (5):
  - Policlinica SelfMed Clinique, Timișoara, Timiș County
  - Sf.Maria Clinical Hospital, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Cluj-Napoca Emergency Clinical County Hospital, Cluj-Napoca
  - Medart Cliniq, Râmnicu Vâlcea
- Spain (4):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital General Universitari de Castello, Castelló
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital de Torrevieja, Torrevieja

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com